CLINICAL TRIAL: NCT06662669
Title: A Randomized, Open, Parallel-controlled, Multi-center , Phase Ib/Ⅱ Clinical Trial of YL-13027 and/or HY-0102 Combined With AG（Nab-paclitaxel and Gemcitabine) Regimen Chemotherapy for Metastatic Pancreatic Cancer
Brief Title: YL-13027 and/or HY-0102 Combined With AG Regimen Chemotherapy for Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YL-13027-004
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Injections; 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GroupA (YL-13027+AG ) (Experimental): YL-13027: 180mg BID PO Nab-paclitaxel: 125mg/m2, ivgtt, D1、D8、D15 Q4W Gemcitabine: 1000mg/m2, ivgtt, D1、D8、D15 Q4W
  Interventions: Drug: YL-13027; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Group B (HY-0102+AG ) (Experimental): HY-0102: 10mg , ivgtt, D1、D15 Q4W Nab-paclitaxel: 125mg/m2, ivgtt, D1、D8、D15 Q4W Gemcitabine: 1000mg/m2, ivgtt, D1、D8、D15 Q4W
  Interventions: Drug: HY-0102; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Group C (YL-13027+HY-0102+AG) (Experimental): YL-13027: 180mg BID PO HY-0102: 10mg , ivgtt, D1、D15 Q4W Nab-paclitaxel: 125mg/m2, ivgtt, D1、D8、D15 Q4W Gemcitabine: 1000mg/m2, ivgtt, D1、D8、D15 Q4W
  Interventions: Drug: YL-13027; Drug: HY-0102; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Group D (AG) (Active Comparator): Nab-paclitaxel: 125mg/m2, ivgtt, D1、D8、D15 Q4W Gemcitabine: 1000mg/m2, ivgtt, D1、D8、D15 Q4W
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: YL-13027 — YL-13027 is a small molecule inhibitor of the TGF-βRI target.
  Other Names: YL-13027 tablet
  Arms: Group C (YL-13027+HY-0102+AG); GroupA (YL-13027+AG )
Drug: HY-0102 — HY-0102 is a recombinant anti-NKG2A humanized monoclonal antibody.
  Other Names: HY-0102 injection
  Arms: Group B (HY-0102+AG ); Group C (YL-13027+HY-0102+AG)
Drug: Gemcitabine — Gemcitabine is a pyrimidine antineoplastic chemotherapeutic agent.
  Other Names: Gemcitabine Hydrochloride for Injection
Drug: Nab-paclitaxel — Paclitaxel for Injection (albumin bound) is a chemotherapeutic agent that acts as an antitumor agent by inhibiting tumor cell mitosis
  Other Names: Paclitaxel for Injection (albumin bound)

SUMMARY:
In Phase 1b study, six subjects will be enrolled in Arm A (YL-13027 + AG regimen) and Arm B (HY-0102 + AG regimen). The first 12 subjects will be evaluated for safety after one cycle. After safety assessment, subjects will start to enroll in Arm C (YL-13027 + HY-0102 + AG regimen). Each group is planned to include 12-20 subjects. According to the safety and efficacy results of 3 arms of subjects in phase Ib, 1-2 groups were selected for expansion, and a randomized controlled study will be conducted with the standard treatment AG （Arm 4）regimen chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 18 and 75 years.
* Subject has histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma.
* Subject has at least one evaluable metastatic lesion according to RECIST 1.1 criteria;
* Subject has an ECOG score of 0-1 and is expected to survive more than 3 months;
* Subjects have a good level of organ function.

Exclusion Criteria:

* Subject suitable for potentially curative surgery.
* The subject confirmed by tissue or cytology as other pathological types, such as acinar cell carcinoma, neuroendocrine carcinoma, etc.
* The subject has previously received gemcitabine and nab-paclitaxel combination therapy within 6 months of progression or intolerance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  The proportion of subjects who have a complete response or partial response.
Progression-free survival | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  Progression-free survival is defined clinically as the time from randomization to disease progression or death from any cause

SECONDARY OUTCOMES:
Disease control rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months.
  The proportion of subjects who have a complete response, partial response and stable disease.
Adverse events | From time of first dose to 30 days after the last dose.
  Incidence of adverse events evaluated by NCI CTCAE v5.0
Plasma concentration of YL-13027 and HY-0102 | From one hour before the first dose to the last dose up to 24months.
  This composite endpoint will measure the plasma concentration of YL-13027 and HY-0102.